CLINICAL TRIAL: NCT01293721
Title: Prospective Randomized Controlled Trial of the Efficacy of Low-Magnitude, High-Frequency Vibration Treatment on Osteoporotic Hip Fracture Healing
Brief Title: Study of Low-Magnitude, High-Frequency Vibration Treatment on Osteoporotic Hip Fracture Healing
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Kwok-Sui Leung, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2008-KSWH
Record Dates: First submitted 2011-02-10; First posted 2011-02-11 (Estimated); Last update posted 2012-05-23 (Estimated); Status verified 2012-05

CONDITIONS: Hip Fracture
Keywords: Bone Mineral Density; Vibration; Rehabilitation; Fracture healing rate
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- control (No Intervention)
- Treatment (Experimental): Receive vibration therapy
  Interventions: Device: Low-magnitude high - frequency vibration treatment

INTERVENTIONS:
Device: Low-magnitude high - frequency vibration treatment — stand on a vibration platform at 35Hz, 0.3g, 20mins/day and 7 days/week
  Arms: Treatment

SUMMARY:
Osteoporotic hip fracture is common in elderly. As a result of aging population in Hong Kong, the total number of hip fracture cases is anticipated to increase substantially in the future, and therefore draw more resources in hospitals and healthcare cost. Osteoporotic hip fracture usually causes severe pain and takes long time (4-8months) to recover due to impaired healing capability in osteoporotic bones and limited mobility. Consequently, the patients will recover very slowly as a result of low physical activities to provide inadequate mechanical stimulation. It is also known that mechanical, vascular and biological factors are the keys for fracture healing.

Low-magnitude, high-frequency vibration (LMHFV) treatment is a biophysical intervention to provide whole-body vibration signals for mechanical stimulation, which has been proven to be good in enhancing bone and muscle performance, as well as blood circulation. Our previous study of LMHFV on femoral fracture in rats showed acceleration of fracture healing, resulted from enhanced callus formation and maturation. Application of LMHFV on osteoporotic fractures could shorten the period of complete callus bridging by 30%. Our clinical trial on normal elderly also demonstrated improved muscle performance with good compliance, which is also a critical factor for fracture healing.

In this study, the investigators therefore hypothesize that LMHFV can enhance hip fracture healing by enhancing fracture impaction, maintaining bone mineral density, enhancing muscle recovery, thus improving implant mechanical stability and rehabilitation in elderly patients. The hip fracture elderly patient will be recruited and randomized into control or treatment group. They will be assessed on the fracture healing at fixed time point. The findings of this study will provide very useful scientific data to support the application of LMHFV for hip fracture patients.The ultimate goal is to enhance the fracture healing and rehabilitation in elderly patients.

ELIGIBILITY:
Inclusion Criteria:

* unilateral hip fracture patients older than 65 years old
* patient fixed with dynamic hip screw

Exclusion Criteria:

* unstable vital signs, large amount of drainage, or wound infection postoperatively
* having of hormone replacement therapy or drug treatment known to affect bone metabolism or cause spontaneous bone loss
* having hypo- or hyperparathyroidism and hypo-, hyperthyroidism, renal or liver disease
* cannot tolerate or complication occurs during study
* patients whose fracture is due to underlying disease, secondary to malignancy

Ages: 65 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 72 (Actual)
Dates: Start 2011-11; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Fracture healing rate | up to 6 months

SECONDARY OUTCOMES:
Balancing ability | second month and sixth month post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kwok Sui Leung, MD, Principal Investigator — Department of Orthopaedics and Traumatology, The Chineses University of Hong Kong
Locations (1):
- Department of Orthopaedics and Traumatology, The Chinese University of Hong Kong, Hong Kong, China